CLINICAL TRIAL: NCT02997878
Title: An Adaptive, Multicentre, Phase IIa, Multi-disease Trial Investigating the Safety & Activity of a Single Infusion of Selected Mesenchymal Stromal Cells in the Treatment of Patients With Primary Sclerosing Cholangitis & Autoimmune Hepatitis
Brief Title: Selected Mesenchymal Stromal Cells to Reduce Inflammation in Patients With PSC and AIH
Acronym: Merlin
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: NHS Blood and Transplant (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG-13-124
Record Dates: First submitted 2016-12-13; First posted 2016-12-20 (Estimated); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Cholangitis, Sclerosing; Hepatitis, Autoimmune
Keywords: Autoimmune; AIH; PSC; Liver disease; Cholangitis
MeSH Terms: conditions — Cholangitis, Sclerosing; Hepatitis, Autoimmune; Liver Diseases; Cholangitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PSC patients (Experimental): Selected Mesenchymal Stromal Cells (dose selection and efficacy) - Orbcel-C. dose selection, combination of 0.5, 1.0,2.5 million cells/kg (3 dose levels). IV single-infusion.
  Interventions: Biological: Orbcel-C
- AIH patients (Experimental): Selected Mesenchymal Stromal Cells (dose selection and efficacy) - Orbcel-C. dose selection, combination of 0.5, 1.0,2.5 million cells/kg (3 dose levels). IV single-infusion.
  Interventions: Biological: Orbcel-C

INTERVENTIONS:
Biological: Orbcel-C — Selected Mesenchymal Stromal Cells derived from human umbilical cord

SUMMARY:
MERLIN is an adaptive, single arm, multi-centre, phase IIa multi-disease clinical trial. It is designed to:

i) Determine dose safety of ORBCEL-C™ (selected Mesenchymal stromal cells derived from human umbilical cord) ii) Evaluate treatment activity through assessment of biomarkers (for patients treated at the highest safe dose only (HSD))

This trial will determine the Highest Safe Dose (HSD) that can be administered by observing for occurrence of dose limiting toxicity (DLT).

Upon completion of this trial we hope to be able to justify and conduct separate, larger scale trials using ORBCEL-C™.

DETAILED DESCRIPTION:
MERLIN is an adaptive, single arm, multi-centre, phase IIa multi-disease clinical trial. It is designed to:

i) Determine dose safety of ORBCEL-C™ (selected Mesenchymal stromal cells derived from human umbilical cord) ii) Evaluate treatment activity through assessment of biomarkers

This trial will determine the HSD* that can be administered by observing for occurrence of dose limiting toxicity (DLT).

* An investigated dose level is determined to be safe if we see 0 DLTs in 3 patients or ((in the instance where a cohort is expanded to 6 patients due to occurrence of a DLT in the first 3 patients treated at a cohort) < 2 DLTs in 6 patients. The HSD is the highest such dose which fulfils these criteria and will be ascertained via dose-escalation using 3+3 methodology.

Further safety and activity outcomes will be determined on patients treated at the HSD only. Upon completion of this trial we hope to be able to justify and conduct separate, larger scale trials using ORBCEL-C™.

OBJECTIVES

For Both Primary Sclerosing Cholangitis (PSC) and Autoimmune Hepatitis (AIH) patients:

The primary objective for all patients is:

• To determine the highest safe single intravenous infusion dose of ORBCEL-C™ over a 14 day (Visit 3 to Visit 5) reporting period.

For patients treated at HSD only, there is an additional co-primary objective:

• To investigate whether a single intravenous infusion of ORBCEL-C™ in patients with PSC and AIH treated at the HSD is safe and tolerated over the period of trial follow-up (up to Visit 8)

For PSC patients only:

• Reduces serum alkaline phosphatase (ALP) in patients with PSC. This is a non- invasive biochemical surrogate of clinical outcomes in PSC

For AIH patients only:

• Reduces serum alanine aminotransferase (ALT) in patients with AIH. This is a non- invasive biochemical surrogate marker of hepatic inflammatory activity and outcomes in AIH.

The secondary objectives are to investigate whether a single intravenous infusion of ORBCEL-C™ elicits a change over the duration of the trial after treatment in all patients with PSC and AIH on:

* Circulating inflammatory cells profile as measured by flow cytometry (key secondary outcome)
* Liver biochemistry and function, immunoglobulin G concentrations (in AIH patients) and composite risk scores
* Non-invasive clinical markers of fibrosis
* Patient Quality of Life (QoL)
* Severity of co-existent Inflammatory Bowel Disease (IBD) in patients with PSC

Further exploratory research objectives of the trial determine whether MSC infusion modulates the immune response by measuring whether treatment elicits a change in all patients with PSC and AIH:

* Markers of immune activation including immunoglobulin values and C-reactive protein (CRP) concentration
* Markers of biliary injury including total bile acid levels
* Endothelial cell activation markers such as VAP-1 and ICAM1
* Serum cytokine, chemokine, ribonucleic acid (RNA) and micro-RNA expression profiles

ELIGIBILITY:
Inclusion Criteria - Patients with Primary Sclerosing Cholangitis (PSC):

1. Age ≥ 18 at Visit 1
2. Diagnosis of PSC at Visit 1 as evidenced clinically by:

   1. Chronic biochemical cholestasis (elevated serum alkaline phosphatase (ALP) above the upper limit of normal (ULN) and/or gamma-glutamyl transpeptidase (GGT) above the ULN) ≥6 months duration AND
   2. Radiological AND/OR histological evidence of clinically documented PSC
3. Serum ALP ≥ 1.5 x ULN at Visit 1
4. Any serum ALP value change is <40% using two sets of laboratory values obtained during screening:

   If a participant fails to confirm an ALP at Visit 2 that is within 40% of the ALP at Visit 1, a further screening ALP (Visit 2a) can be arranged, so long as the variation in ALP was <50%, and the Principal Investigator has no other clinical reason to suggest the participant is clinically unstable. If the ALP is within 40% variance at Visit 2a as compared to visit 1, Trial registration is permitted.
5. At Visit 2 (and Visit 2a if applicable), it should be confirmed that a patient does not meet any of the exclusion criteria

Inclusion Criteria - Patients with Autoimmune Hepatitis (AIH):

1. Age ≥ 18 at Visit 1
2. Established pre-existing clinical diagnosis of AIH confirmed by clinical expert review consistent with the simplified IAIHG criteria (http://www.mdcalc.com/simplified-scoring-autoimmune-hepatitis-aih/) and must include history of a liver biopsy reported compatible with AIH
3. Active AIH defined by ALT ≥ 1.1 x ULN
4. Serum ALT must be above ≥ 1.1 x ULN at both Visit 1 and Visit 2
5. At Visit 2, it should be confirmed that a patient does not meet any of the exclusion criteria
6. Patients must be on standard-of-care AIH treatment for ≥ 24 weeks -this includes any AIH therapy except biologics
7. Stable doses of immunosuppression for a minimum period of 4 weeks (28 days) at the time of Visit 1.

Exclusion Criteria - Patients with PSC and AIH:

Patients who meet any of the following exclusion criteria are excluded from participating in the MERLIN trial

1. Refusal or lacks capacity to give informed consent to participate in trial
2. Patient who is unable to participate in follow-up assessment
3. Participation actively, or within 5 half-lives, of another interventional clinical trial
4. Known hypersensitivity to the investigational product or any of its formulation excipients
5. Evidence of active malignancy (within 3 years of Visit 1), other than non-melanomatous skin cancer and cervical dysplasia in situ
6. Major surgical procedure within 30 days at Visit 1
7. Prior organ transplantation
8. Active harmful alcohol consumption as evaluated and documented by the Investigator
9. Poor venous access, therefore unable to support a 22G needle for infusion
10. Creatinine > 133 μmol/L or being treated with renal replacement therapy at the time of Visit 1
11. AST or ALT > 10 x ULN
12. ALP > 10 x ULN
13. Platelets < 50 x 10^9/L
14. Total Bilirubin > 2 x ULN
15. INR > 1.3 (in the absence of concomitant use of Warfarin or equivalent anti-coagulant therapy)
16. Albumin < 35 g/L
17. Haemoglobin < 10 g/dL
18. Past or present evidence of decompensated chronic liver disease:

    1. Radiological or clinical evidence of ascites
    2. Hepatic encephalopathy
    3. Endoscopic evidence for portal hypertensive bleeding
19. Any active treatment with biologic therapy (monoclonal antibodies)
20. Clinically severe cardiovascular disease as evaluated by the Investigator
21. Pregnancy or breast-feeding
22. Women of child bearing potential who are unwilling to practice effective contraception (i.e. barrier, oral contraceptive pill, implanted contraception, or previous hysterectomy, bilateral oophorectomy) for the duration of the trial up to 90 days after the trial drug is administered. If using hormonal agents the same method must have been used for at least 1 month before trial dosing and patients must use a barrier method during that time period
23. Non-vasectomised men, sexually active with women of child bearing potential, who are not willing to practice effective contraception (condom with spermicide) for the duration of the trial up to 90 days after the trial drug is administered
24. Patients with a history of hepatitis C (present or past infection), known positivity for antibody to HIV or any evidence of current or past hepatitis B infection
25. Presence of an acute/chronic infection or illness that, at the discretion of the Investigator, might compromise the patient's health and safety in the trial
26. Any symptoms indicative of Covid-19; including fever, chronic/persistent cough, or loss of sense of taste or smell in the preceding two weeks.
27. Receipt of live vaccination within six weeks prior to Visit 1

Exclusion Criteria Specific to Patients with PSC:

1. Documented alternative aetiology for sclerosing cholangitis (i.e. secondary sclerosing cholangitis)
2. A dominant (as determined by Investigator) alternative chronic or active liver injury other than PSC at the time of Visit 1; Patients with possible overlap syndrome with AIH are excluded from the PSC cohort if the Investigator considers AIH as the dominant liver injury
3. UDCA dose modification within the last 90 days
4. ALP > 10 x ULN
5. Evidence of cholangitis within 90 days of Visit 1

   1. Documented evidence of cholangitis by physician
   2. Need for any antibiotics for presumed cholangitis
6. Any patient taking prophylactic antibiotics to combat recurrent cholangitis
7. Presence of percutaneous biliary drain, or internal biliary stent
8. Diagnosed hepatocellular carcinoma or cholangiocarcinoma or high clinical suspicion thereof
9. Dominant stricture clinically suspicious of cholangiocarcinoma (as determined by Investigator)

Exclusion Criteria for PSC patients with IBD:

1. Unstable disease as evidenced by:

   1. Documented clinically significant flare within 90 days of enrolment requiring any marked intensification of therapy from baseline maintenance (maintenance therapy = thiopurines, 5- aminosalicylates, or oral prednisolone < 10mg/day; biologics therapy is an exclusion criteria
   2. Requirement for daily prednisolone > 10mg
   3. Mayo Clinic Score ≥ 2 (see Appendix 1 for details) AND clinician assessment of active disease requiring up-titration of treatment; last colonoscopy within last year used for endoscopic component
2. Any colonoscopic evidence of clinically significant dysplasia at last colonoscopy
3. Patients who have not had their routine colonoscopy within 24 months prior to planned MSC infusion and are unable to have their screening colonoscopy examination as per standard care prior to Visit 3
4. A Mayo score/ Disease Activity Index for Ulcerative Colitis of ≥ 5 (https://www.mdcalc.com/mayo-score- disease-activity-index-dai-ulcerative-colitis)

Exclusion Criteria Specific to Patients with AIH:

1. A dominant (as determined by Investigator) alternative chronic or active liver injury other than AIH at the time of Visit 1; Patients with possible overlap syndrome with PSC are excluded from the AIH cohort if the Investigator considers PSC as the dominant liver injury
2. AST or ALT > 10 x ULN
3. Patients on a prednisolone dose of > 20 mg at the time of screening
4. Treatment with biologic therapy within 24 weeks of the time of screening
5. Patients with a history of poor compliance with medication
6. Diagnosed hepatocellular carcinoma or cholangiocarcinoma or high clinical suspicion thereof

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-12-07 (Actual); Primary Completion 2023-11-23 (Actual); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Dose finding and incidence of treatment emergent adverse events (safety and tolerability) in all PSC and AIH Patients | Visit 3 to Visit 5 -14 days
  Occurrence of Dose Limiting Toxicity (DLT) over 14 day (Visit 3 to Visit 5) reporting period after ORBCEL-C infusion
Incidence of treatment emergent adverse events (safety and tolerability) for PSC and AIH patients treated at the Highest Safe Dose (HSD) only | Visit 3 to Visit 8 - 56 days
  Determine safety and tolerability by occurrence of Dose Limiting Toxicity (DLT) (Visit 3 to Visit 5 only), Serious Adverse Events (SAEs) and Adverse Events (AEs) throughout trial period (up to Visit 8)
Activity and Safety at the Highest Safe Dose (HSD) of ORBCEL-C in PSC patients, by measure of change in Alkaline Phosphatase (ALP) | Baseline to Visit 8 - Approximately 80 days
  Change in Alkaline Phosphatase (ALP) after ORBCEL-C infusion - Examination of change in ALP at Day 28 from Baseline and changes over multiple time-points before and after infusion (Visit 1 to Visit 8)
Activity at the Highest Safe Dose (HSD) of ORBCEL-C in AIH patients, by measure of change in Alanine Aminotransferase (ALT) | Baseline to Visit 8 - Approximately 80 days
  Change in Alanine Aminotransferase (ALT) trend after ORBCEL-C infusion. Measurements of ALT will be taken at multiple time points from Visit 1 to Visit 8.

SECONDARY OUTCOMES:
All patients with Autoimmune Hepatitis (AIH) - Secondary Outcome Measure 1 | Baseline to Visit 8 - Approximately 80 days
  Change from baseline at Visit 7, Visit 8 and throughout the trial period (up to Visit 8) following ORBCEL-C™ infusion in Phenotypic expression of TRegs as measured by flow cytometry (principal secondary outcome)
All patients with Autoimmune Hepatitis (AIH) - Secondary Outcome Measure 2 | Baseline to Visit 8 - Approximately 80 days
  Change from baseline at Visit 7, Visit 8 and throughout the trial period (up to Visit 8) following ORBCEL-C™ infusion in Individual markers of liver biochemistry and function including AST, ALP, GGT, bilirubin, albumin, INR and composite risk score (MELD)
All patients with Autoimmune Hepatitis (AIH) - Secondary Outcome Measure 3 | Baseline to Visit 8 - Approximately 80 days
  Change from baseline at Visit 7, Visit 8 and throughout the trial period (up to Visit 8) following ORBCEL-C™ infusion in marker of immune activation - immunoglobulin G concentrations
All patients with Autoimmune Hepatitis (AIH) - Secondary Outcome Measure 4 | Baseline to Visit 8 - Approximately 80 days
  Change from baseline at Visit 7, Visit 8 and throughout the trial period (up to Visit 8) following ORBCEL-C™ infusion in Non-invasive clinical markers of fibrosis - ELF and transient elastography (Fibroscan®)
All patients with Autoimmune Hepatitis (AIH) - Secondary Outcome Measure 5 | Baseline to Visit 8 - Approximately 80 days
  Change from baseline at Visit 7, Visit 8 and throughout the trial period (up to Visit 8) following ORBCEL-C™ infusion in QoL as measured by Pruritus Visual Analogue Scale, nine-point fatigue severity scale and SF-36v2
All patients with Primary Sclerosing Cholangitis (PSC) - Secondary Outcome Measure 1 | Baseline to Visit 8 - Approximately 80 days
  Change from baseline at Visit 7, Visit 8 and throughout the trial period (up to Visit 8) following ORBCEL-C™ infusion in Phenotypic expression of TRegs as measured by flow cytometry (principal secondary outcome)
All patients with Primary Sclerosing Cholangitis (PSC) - Secondary Outcome Measure 2 | Baseline to Visit 8 - Approximately 80 days
  Change from baseline at Visit 7, Visit 8 and throughout the trial period (up to Visit 8) following ORBCEL-C™ infusion in Individual markers of liver biochemistry and function including aspartate aminotransferase (AST), alanine transaminase (ALT), gamma-glutamyl transpeptidase (GGT), bilirubin, albumin, international normalised ratio [INR] and composite risk scores (Mayo PSC risk score and Model for End Stage Liver Disease [MELD])
All patients with Primary Sclerosing Cholangitis (PSC) - Secondary Outcome Measure 3 | Baseline to Visit 8 - Approximately 80 days
  Change from baseline at Visit 7, Visit 8 and throughout the trial period (up to Visit 8) following ORBCEL-C™ infusion in Non-invasive clinical markers of fibrosis: Enhanced Liver Fibrosis (ELF) and transient elastography (Fibroscan®)
All patients with Primary Sclerosing Cholangitis (PSC) - Secondary Outcome Measure 4 | Baseline to Visit 8 - Approximately 80 days
  Change from baseline at Visit 7, Visit 8 and throughout the trial period (up to Visit 8) following ORBCEL-C™ infusion in QoL as measured by Pruritus Visual Analogue Scale, nine-point fatigue severity scale and SF-36v2 Severity of IBD as measured by the non-endoscopic aspects of the Mayo IBD score - stool frequency, rectal bleeding, and physician's global assessment

OTHER OUTCOMES:
All patients with PSC and AIH - Exploratory Research Outcome 1 | Up to Visit 8 (56 days)
  Change throughout the trial period up to Visit 8 of the following measured parameters:
  Markers of immune activation including immunoglobulin values and C-reactive protein concentration
All patients with PSC and AIH - Exploratory Research Outcome 2 | Up to Visit 8 (56 days)
  Change throughout the trial period up to Visit 8 of the following measured parameters: Markers of biliary injury including total bile acid levels (these will only be measured prior to infusion at Visit 3 and Visit 7)
All patients with PSC and AIH - Exploratory Research Outcome 3 | Up to Visit 8 (56 days)
  Change throughout the trial period up to Visit 8 of the following measured parameters: Circulating inflammatory cells profile as measured by flow cytometry Endothelial cell activation markers such as VAP-1 and ICAM1
All patients with PSC and AIH - Exploratory Research Outcome 4 | Up to Visit 8 (56 days)
  Change throughout the trial period up to Visit 8 of the following measured parameters: Serum cytokine and chemokine profiles as measured by cytokine array analysis
All patients with PSC and AIH - Exploratory Research Outcome 5 | Up to Visit 8 (56 days)
  Change throughout the trial period up to Visit 8 of the following measured parameters: RNA and micro-RNA profiles in circulating cells as measured by quantitative polymerase chain reaction (qPCR) or equivalent technology

CONTACTS AND LOCATIONS:
Overall Officials: Phillip N Newsome, Prof, Principal Investigator — University of Birmingham
Locations (1):
- University Hospitals Birmingham NHS Foundation Trust, Queen Elizabeth Hospital, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No